CLINICAL TRIAL: NCT02622438
Title: Course and Follow up of Patients Affected by Facioscapulohumeral Muscular Dystrophy
Brief Title: Routine Health Care of Patients With FSHD
Acronym: FSHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9371
Record Dates: First submitted 2015-11-30; First posted 2015-12-04 (Estimated); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Primary Disease Fascioscapulohumeral Dystrophy (FSHD)
Keywords: FSHD; Usual care performed at Montpellier hospital; Muscle function; Antioxidants; Oxidative stress; Quality of life; Physical activities, development of food-based dietary guidelines; Co-morbidity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Course and follow up of patients affected by FSHD (Other)
  Interventions: Other: Followed with an initial assessment, 12 months and followed annually corresponding to the usual follow-up of the patient.

INTERVENTIONS:
Other: Followed with an initial assessment, 12 months and followed annually corresponding to the usual follow-up of the patient.

SUMMARY:
On the basis of published data and our results indicating that oxidative stress may contribute to the peripheral skeletal muscle dysfunction in patients with FSHD, investigators conducted a pilot randomized double-blind placebo controlled trial to test whether oral administration of vitamins and mineral could improve the physical performance of patients with FSHD.The result of this clinical trial showed that antioxidants supplementation may improve skeletal muscle function of patients with FSHD and suggest that an antioxidant strategy adapted may be a relevant therapeutic approach for these patients. Since then, patients with FSHD who attend consultation at Montpellier hospital are systematically supplemented with antioxidants according their own blood tests.

DETAILED DESCRIPTION:
This study will assess course of patients with FSHD in accordance with usual care performed within the Department of clinical physiology at the University hospital of Montpellier. This prospective longitudinal study include an initial assessment. Then the follow up of patients will be monitored at 12 months and annually. The eventual objective will be to develop a FSHD disease cohort in care at the Montpellier hospital. A statistical analysis will be performed at 3-years follow-up

ELIGIBILITY:
Inclusion Criteria:

* Molecular and clinical diagnosis for FSHD
* patients, men and women aged > 7 years,

Exclusion Criteria:

* pregnant women
* Inability to understand the nature and goals of the study and / or communication difficulties with the investigator
* Major protected by law (guardianship, curatorship or under judicial protection)

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-04-19 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Effect of usual care performed at Montpellier hospital on the measurement of the maximal voluntary contraction (MVC) of quadriceps expressed in kg | 1 day (the day of inclusion)
Effect of usual care performed at Montpellier hospital on the measurement of the maximal voluntary contraction (MVC) of quadriceps expressed in kg | 12 months after inclusion
Effect of usual care performed at Montpellier hospital on the measurement of the maximal voluntary contraction (MVC) of quadriceps expressed in kg | 24 months after inclusion
Effect of usual care performed at Montpellier hospital on the measurement of the maximal voluntary contraction (MVC) of quadriceps expressed in kg | 36 months after inclusion
Effect of usual care performed at Montpellier hospital on the measurement of the maximal voluntary contraction (MVC) of quadriceps expressed in kg | 48 months after inclusion
Effect of usual care performed at Montpellier hospital on the measurement of the maximal voluntary contraction (MVC) of quadriceps expressed in kg | 60 months after inclusion

SECONDARY OUTCOMES:
Effect of usual care performed at Montpellier hospital on quality of life (SF36 questionnaire) | 1 day (the day of inclusion)
Effect of usual care performed at Montpellier hospital on quality of life (SF36 questionnaire) | 12 months after inclusion
Effect of usual care performed at Montpellier hospital on quality of life (SF36 questionnaire) | 24 months after inclusion
Effect of usual care performed at Montpellier hospital on quality of life (SF36 questionnaire) | 36 months after inclusion
Effect of usual care performed at Montpellier hospital on quality of life (SF36 questionnaire) | 48 months after inclusion
Effect of usual care performed at Montpellier hospital on quality of life (SF36 questionnaire) | 60 months after inclusion
Effect of usual care performed at Montpelier hospital on physical activities (Vorrips questionnaire) | 1 day (the day of inclusion)
Effect of usual care performed at Montpellier hospital on physical activities (Vorrips questionnaire) | 12 months after inclusion
Effect of usual care performed at Montpelier hospital on physical activities (Vorrips questionnaire) | 24 months after inclusion
Effect of usual care performed at Montpelier hospital on physical activities (Vorrips questionnaire) | 36 months after inclusion
Effect of usual care performed at Montpelier hospital on physical activities (Vorrips questionnaire) | 48 months after inclusion
Effect of usual care performed at Montpelier hospital on physical activities (Vorrips questionnaire) | 60 months after inclusion
Effect of usual care performed at Montpellier hospital on oxidative stress markers measured by laboratory tests | 1 day (the day of inclusion)
Effect of usual care performed at Montpellier hospital on oxidative stress markers measured by laboratory tests | 12 months after inclusion
Effect of usual care performed at Montpellier hospital on oxidative stress markers measured by laboratory tests | 24 months after inclusion
Effect of usual care performed at Montpellier hospital on oxidative stress markers measured by laboratory tests | 36 months after inclusion
Effect of usual care performed at Montpellier hospital on oxidative stress markers measured by laboratory tests | 48 months after inclusion
Effect of usual care performed at Montpellier hospital on oxidative stress markers measured by laboratory tests | 60 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jacques MERCIER, MD PhD, Principal Investigator — CHRU de Montpellier
Locations (1):
- Montpellier University Hospital- Saint Eloi Hospital, Montpellier, Languedoc-Roussillon, France